CLINICAL TRIAL: NCT04153188
Title: Pilot Study to Evaluate Vbeam® Prima Pulsed Dye Laser (PDL) Treatment and RHOFADE® (Oxymetazoline HCL, 1% Cream) for Erythematotelangiectatic Rosacea
Brief Title: Pulsed Dye Laser Treatment and Oxymetazoline Hydrochloride (HCL) 1% Cream for Erythematotelangiectatic Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHF24671
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: Erythema; Rosacea; Telangiectasia; pulsed dye laser; oxymetazoline hydrochloride 1% cream
MeSH Terms: conditions — Rosacea; Erythema; Telangiectasis | interventions — Oxymetazoline

STUDY DESIGN:
Intervention Model Description: Subjects randomized at baseline to either 3 monthly treatments with PDL and daily oxymetazoline 1.0% cream (Arm 1) or oxymetazoline cream alone (Arm 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pulsed Dye Laser & Oxymetazoline HCL 1% Cream (Experimental): Once daily application of pea-sized amount to face of Oxymetazoline HCL 1% Cream for 4 weeks prior to 1st of 3 monthly Vbeam® Prima PDL treatments. Subjects will continue with once daily application of Oxymetazoline HCL 1% Cream during the 6-month post-baseline study with a 3-day washout of cream prior to each of the 3 PDL treatments.
  Interventions: Device: The Vbeam® Prima System; Drug: Oxymetazoline HCL 1% Cream
- Oxymetazoline HCL 1% Cream (Active Comparator): Once daily application of pea-sized amount to face of Oxymetazoline HCL 1% Cream during the 6-month study.
  Interventions: Drug: Oxymetazoline HCL 1% Cream

INTERVENTIONS:
Device: The Vbeam® Prima System — 3 monthly Vbeam® Prima PDL treatments with a 3-day washout of topical Oxymetazoline HCL 1% cream before each treatment.
  Other Names: Vbeam® Prima Pulsed Dye Laser Treatment; Pulsed Dye Laser Treatment; PDL Treatment
  Arms: Pulsed Dye Laser & Oxymetazoline HCL 1% Cream
Drug: Oxymetazoline HCL 1% Cream — Daily application of Oxymetazoline HCL 1% cream for the 6-month study.
  Other Names: RHOFADE®

SUMMARY:
This study will compare treatment outcome with pulsed dye laser, when used used as an adjunctive treatment to oxymetazoline HCl 1% cream, compared to oxymetazoline HCL 1% cream alone, for patients with moderate or severe erythematotelangiectatic rosacea.

DETAILED DESCRIPTION:
This is a prospective, two-arm randomized, baseline-controlled, pilot study to evaluate treatment outcome of 3 Vbeam® Prima PDL treatments in subjects applying once-daily RHOFADE® topical oxymetazoline HCL 1.0% cream for improvement in erythematotelangiectatic rosacea. Treatment outcome will be compared to oxymetazoline HCL 1% cream alone.

Subjects with moderate or severe (Grade 3 or 4) erythematotelangiectatic rosacea on the validated Clinical Erythema Assessment (CEA) Scale and Subject Self-Assessment (SSA) Scale will be enrolled and randomized to one of two study arms:

Arm 1- 3 monthly treatments with Vbeam® PDL with daily RHOFADE® topical oxymetazoline HCL 1.0% cream.

Arm 2 -Treatment with daily RHOFADE® topical oxymetazoline HCL 1.0% cream only.

All subjects will apply RHOFADE® cream daily during the 6-month study. After 1-month of RHOFADE® cream, subjects in the combined treatment Arm 1 will receive the first of three monthly Vbeam® PDL treatments (at 4-week intervals) with a 3-day washout of cream before each treatment.

Investigators will assess erythema severity, global aesthetic improvement and vessel size improvement with treatment at 1, 2, 3 and 6-months' post-baseline. Subject satisfaction will be assessed. Safety assessments will be conducted at each study visit, and subjects in Arm 1 will also be assessed for treatment-associated discomfort and post-treatment response following PDL treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male or female of 18 to 75 years of age.
2. Subject has erythematotelangiectatic rosacea with clinician erythema assessment (CEA) and subject self-assessment (SSA) of "moderate" or "severe" (Grade 3 or 4).
3. Fitzpatrick Skin Type I - VI.
4. Subject must be able to read, understand and sign the Informed Consent Form.
5. Subject must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
6. Subject must be willing to have limited sun exposure for the duration of the study, including the follow-up period up to 6 months post-baseline.
7. Subject is willing to have photographs taken of the treated area that will be used, de-identified, in evaluations and may be used, de-identified, in presentations and/or publications.
8. For female candidates - subject must be post-menopausal, or surgically sterilized, or using a medically acceptable form of birth control during the entire course of the study.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant during the study duration.
2. Subject has an active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Subject has an implant in the treated area (such as metal plates or screws) or an injected chemical substance.
4. Subject has a known collagen (connective tissue) disorder, vascular disease, scleroderma or other autoimmune disease (i.e. rheumatoid arthritis, lupus).
5. Subject has a history of diseases stimulated by heat or sun exposure, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
6. Subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
7. Having or undergoing any form of treatment for active cancer or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
8. Subject is suffering from significant concurrent illness, such as such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
9. Subject has an infection or is suffering from current or has a history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: photodermatoses, active acne, excessive skin dryness, psoriasis, eczema, rash, open wounds, varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
10. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use might be requested as per the subject's physician discretion).
11. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session.
12. Subject has a history of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
13. Subject has a history of keloid scarring or of abnormal wound healing.
14. Subject has a known photosensitivity to the device's laser wavelengths, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
15. Subject has undergone any surgical, light-based therapy or radiofrequency (RF) procedures in the treatment area within 3 months of treatment or during the study.
16. Having undergone any other surgery in the treated area within 3 months of treatment (or more if skin has not healed completely) or during the study.
17. Subject has a tattoo or permanent make-up in the treated area.
18. Subject has systemically used retinoids or antioxidants within 1 month of treatment or during the study.
19. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
20. Participation in a study of another device or drug within three months prior to enrollment or during the study.
21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konika P Schallen, MD, Study Director — Candela Corporation
Locations (2):
- United States (2):
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Dermatology & Laser Surgery Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan J, Liu H, Leyden JJ, Leoni MJ. Reliability of Clinician Erythema Assessment grading scale. J Am Acad Dermatol. 2014 Oct;71(4):760-3. doi: 10.1016/j.jaad.2014.05.044. Epub 2014 Jul 4. PMID 24999270
- [Background] DuBois J, Dover JS, Jones TM, Weiss RA, Berk DR, Ahluwalia G. Phase 2 Randomized, Dose-Ranging Study of Oxymetazoline Cream for Treatment of Persistent Facial Erythema Associated With Rosacea. J Drugs Dermatol. 2018 Mar 1;17(3):308-316. PMID 29537449
- [Background] Bernstein EF, Schomacker K, Paranjape A, Jones CJ. Pulsed dye laser treatment of rosacea using a novel 15 mm diameter treatment beam. Lasers Surg Med. 2018 Oct;50(8):808-812. doi: 10.1002/lsm.22819. Epub 2018 Apr 10. PMID 29635699
- [Background] Suggs AK, Macri A, Richmond H, Munavalli G, Friedman PM. Treatment of Erythematotelangiectatic Rosacea With Pulsed-Dye Laser and Oxymetazoline 1.0% Cream: A Retrospective Study. Lasers Surg Med. 2020 Jan;52(1):38-43. doi: 10.1002/lsm.23176. Epub 2019 Nov 10. PMID 31709571
- [Result] Sodha P, Suggs A, Munavalli GS, Friedman PM. A Randomized Controlled Pilot Study: Combined 595-nm Pulsed Dye Laser Treatment and Oxymetazoline Hydrochloride Topical Cream Superior to Oxymetazoline Hydrochloride Cream for Erythematotelangiectatic Rosacea. Lasers Surg Med. 2021 Dec;53(10):1307-1315. doi: 10.1002/lsm.23439. Epub 2021 Jul 7. PMID 34233378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each subject was randomly assigned to receive either oxymetazoline therapy combined with three monthly 595-nm PDL treatments (Arm 1) or oxymetazoline therapy only (Arm 2). Accordingly, eighteen subjects were assigned to Arm 1 and sixteen subjects were assigned to Arm 2.
Pre-assignment Details: Four subjects dropped prior to 1 month post baseline visit (three subjects from Arm 2 and one subject from Arm 1). Therefore, thirty subjects are included in the analysis (17 subjects from Arm 1 and 13 subjects from Arm 2)
Period: Overall Study
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Started | 17 | 13
Completed | 14 | 11
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subject withdrew due to rebound erythema when Oxymetazoline wore off | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 46 (9) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 12 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 12 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30
Clinical Erythema Assessment (CEA) Score [Mean (Standard Deviation); unit: units on a scale] — Investigator Clinical Erythema Assessment (CEA): A five category scale ranging from 0 [clear skin with no signs of erythema] to 4 [severe erythema; fiery redness]
  units on a scale | 3.2 (0.4) | 3.2 (0.4) | 3.2 (0.4)
Subject Self-Assessment [Mean (Standard Deviation); unit: units on a scale] — Subject Self-Assessment (SSA): A five category scale ranging from 0 [Clear of unwanted redness] to 4 [Completely unacceptable redness].
  units on a scale | 3.5 (0.5) | 3.6 (0.5) | 3.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Erythema Assessment (CEA) Score At 6-Month Post-Baseline
Description: CEA was graded by the investigator according to 5-point scale (0=Clear to 4=Severe) for each patient at the 6-month post-baseline visits. A higher score indicates worse outcome. The outcomes presented here are the mean CEA calculated for the 6-month post-baseline visit of each arm.
Time Frame: 6-month post-baseline
Population: Arm 1- Two subjects dropped before 2-month post-baseline visit and one subject dropped before the 6-month post baseline visit.
  Arm 2- One subject dropped before 2-month post-baseline visit and one subject dropped before the 6-month post baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 14 | 11
score on a scale | 1.6 (1.0) | 2.4 (1.0)

2. Secondary Outcome: Clinical Erythema Assessment (CEA) At the 1- ,2- and 3-Month Post-Baseline Visits
Description: Clinical Erythema Assessment (CEA) scores at the 1- ,2- and 3-month post-baseline visits were assessed for each patient by the investigator. CEA scores were graded according to 5-point scale (0=Clear to 4=Severe). A higher score indicates worse outcome. The outcomes presented here are the mean CEA calculated for each visit.
Time Frame: 1- ,2- and 3-Month Post-Baseline Visits
Population: Arm 1- Two subjects dropped before 2-month post-baseline visit. Arm 2- One subject dropped before 2-month post-baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17 | 13
score on a scale
  Clinical Erythema Assessment (CEA) At 1-Month Post-Baseline | 2.6 (0.8) | 2.6 (0.5)
  Clinical Erythema Assessment (CEA) At 2-Month Post-Baseline: number analyzed (Participants) | 15 | 12
  Clinical Erythema Assessment (CEA) At 2-Month Post-Baseline | 2.5 (0.6) | 2.0 (0.6)
  Clinical Erythema Assessment (CEA) At 3-Month Post-Baseline: number analyzed (Participants) | 15 | 12
  Clinical Erythema Assessment (CEA) At 3-Month Post-Baseline | 2.0 (0.8) | 2.3 (0.8)

3. Secondary Outcome: Subject Self-Assessment (SSA) At the 1- ,2-, 3- and 6-Month Post-Baseline Visits
Description: Subject Self-Assessment (SSA) at the 1- ,2-, 3- and 6-month post-baseline visits were graded according to 5-point scale (0=Clear of unwanted redness to 4=Completely unacceptable redness) at each visit. A higher score indicates worse outcome.
Time Frame: 1-, 2-, 3- and 6-months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17 | 13
score on a scale
  Subject Self-Assessment (SSA) At the 1-Month Post Baseline | 3.3 (0.8) | 3.0 (0.6)
  Subject Self-Assessment (SSA) At the 2-Month Post Baseline: number analyzed (Participants) | 15 | 12
  Subject Self-Assessment (SSA) At the 2-Month Post Baseline | 2.7 (1.0) | 2.3 (0.7)
  Subject Self-Assessment (SSA) At the 3-Month Post Baseline: number analyzed (Participants) | 15 | 12
  Subject Self-Assessment (SSA) At the 3-Month Post Baseline | 2.1 (1.1) | 2.3 (0.7)
  Subject Self-Assessment (SSA) At the 6-Month Post Baseline: number analyzed (Participants) | 14 | 11
  Subject Self-Assessment (SSA) At the 6-Month Post Baseline | 1.4 (1.2) | 2.2 (0.9)

4. Secondary Outcome: Mean Investigator Assessment of Global Aesthetic Improvement (GAI) Grades At the 1-, 2-, 3- and 6-Month Post-Baseline
Description: Investigator measurement of Global Aesthetic Improvement (GAI) with treatment. GAI is graded according to 5-point scale (0=Excellent improvement to 4=No change). A higher score indicates a worse outcome. The outcomes presented here are the mean GAI calculated for each visit.
Time Frame: 1-, 2-, 3- and 6-month post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17 | 13
score on a scale
  Mean GAI Grade at 1-Months Post-Baseline Visit | 2.5 (1.2) | 2.7 (1.0)
  Mean GAI Grade at 2-Months Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean GAI Grade at 2-Months Post-Baseline Visit | 2.3 (1.1) | 1.4 (1.0)
  Mean GAI Grade at 3-Months Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean GAI Grade at 3-Months Post-Baseline Visit | 1.7 (1.4) | 2.5 (1.6)
  Mean GAI Grade at 6-Months Post-Baseline Visit: number analyzed (Participants) | 14 | 11
  Mean GAI Grade at 6-Months Post-Baseline Visit | 1.2 (1.4) | 2.5 (1.3)

5. Secondary Outcome: Mean Subject Assessment of Global Aesthetic Improvement (GAI) Grades At the 1-, 2-, 3- and 6-Month Post-Baseline
Description: Subject measurement of Global Aesthetic Improvement (GAI) with treatment. GAI is graded according to 5-point scale (0=Excellent improvement to 4=No change). A higher score indicates a worse outcome. The outcomes presented here are the mean GAI calculated for each visit.
Time Frame: 1-, 2-, 3- and 6-month post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17 | 13
units on a scale
  Mean GAI Grade at 1-Months Post-Baseline Visit | 2.6 (1.0) | 2.9 (1.0)
  Mean GAI Grade at 2-Months Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean GAI Grade at 2-Months Post-Baseline Visit | 1.9 (0.8) | 2.4 (0.7)
  Mean GAI Grade at 3-Months Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean GAI Grade at 3-Months Post-Baseline Visit | 1.2 (1.0) | 2.6 (0.9)
  Mean GAI Grade at 6-Months Post-Baseline Visit: number analyzed (Participants) | 14 | 11
  Mean GAI Grade at 6-Months Post-Baseline Visit | 0.7 (0.9) | 2.1 (0.9)

6. Secondary Outcome: Measurement of Improvement in Vessel Size At the 1-, 2-, 3- and 6-Month Post-Baseline Visits
Description: Investigator assessment of improvement in vessel size with treatment. Improvement in vessel size is graded according to 4-point scale (0=76-100% improvement (excellent) to 4=No response). A higher score indicates a worse outcome. Mean score was calculated for each visit.
Time Frame: 1-, 2-, 3- and 6-month post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17 | 13
score on a scale
  Mean Vessel Size Improvement Grade at 1-Month Post-Baseline Visit | 3.4 (0.9) | 3.2 (0.7)
  Mean Vessel Size Improvement Grade at 2-Month Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean Vessel Size Improvement Grade at 2-Month Post-Baseline Visit | 2.4 (1) | 2.7 (1.1)
  Mean Vessel Size Improvement Grade at 3-Month Post-Baseline Visit: number analyzed (Participants) | 15 | 12
  Mean Vessel Size Improvement Grade at 3-Month Post-Baseline Visit | 1.8 (1.1) | 3.1 (1.2)
  Mean Vessel Size Improvement Grade at 6-Month Post-Baseline Visit: number analyzed (Participants) | 14 | 11
  Mean Vessel Size Improvement Grade at 6-Month Post-Baseline Visit | 1.6 (1.5) | 3.1 (0.9)

7. Secondary Outcome: Measurement of The Percentage of Subjects Reporting Satisfaction At the 6-Month Post-Baseline Visit
Description: Subject satisfaction is graded according to 5-point scale (0=Very Satisfied to 4=Very Dissatisfied). Lower score indicates higher satisfaction. A score of 0 or 1 indicates satisfaction with treatment outcome. The measurements reflect the percentage of subjects that were satisfied (graded 0 or 1) at the 6-month post-baseline visit
Time Frame: 6-month post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 14 | 11
Participants | 12 | 7

8. Secondary Outcome: Measurement of Pain Associated With PDL Treatment
Description: A standard 10-centimeter visual analog scale from 0=No pain to 10=worst pain was used by subjects to report pain level associated with PDL treatment. A higher score indicates greater pain/discomfort with treatment. Mean of all pain associated scores obtained for all PDL treatments was calculated.
Time Frame: 1-, 2- and 3-month post-baseline
Population: Arm 1- Two subjects dropped before 2-month post-baseline visit. Therefore 17 subjects underwent the first treatment and 15 subjects underwent a second and third treatments.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: PDL Treatments
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream
Number analyzed (Participants) | 17
Number analyzed (PDL Treatments) | 47
score on a scale | 4.5 (2.2)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected is from first visit until 6 month post baseline
Description: The number and severity of adverse events following Oxymetazoline and/or Pulsed Dye Laser treatments for Arm 1 (Pulsed Dye Laser & Oxymetazoline HCL 1 % Cream) or following Oxymetazoline treatment for Arm 2 (Oxymetazoline HCL 1 % Cream). Adverse events were evaluated at each of the visits following baseline until the last visit (6 month post baseline).
Arm/Group | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream | Oxymetazoline HCL 1% Cream
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 3/17 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Dye Laser & Oxymetazoline HCL 1% Cream (N=17) | Oxymetazoline HCL 1% Cream (N=13)
Dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Mild dryness from oxymetazoline usage on the cheeks and forehead reported at the 1 month post baseline visit - 1 experienced at the first week of usage - both adverse events recovered without intervention before the 1 month post baseline visit.
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Subject experienced mild tingling sensation on the cheeks after applying oxymetazoline, but improved after continued use.
Blistering (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Mild blistering that appeared on the skin after first PDL treatment. Both cases resolved spontaneously before the 1-week post treatment visit.
Edema and Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild case of prolong edema and erythema on the cheeks and forehead after the first PDL treatment that has recovered without intervention after the 1-week follow up
Papules (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Papules on the cheeks and forehead within the first month of oxymetazoline cream, which improved after several weeks of applying topical SOOLANTRA ® (ivermectin) cream, 1%.

LIMITATIONS AND CAVEATS:
Small sample size for randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04153188/Prot_SAP_000.pdf